CLINICAL TRIAL: NCT06404840
Title: Evaluating Nimotuzumab in Combination With AG Regimen for Pancreatic Cancer With Liver Metastases (PCLM): A Prospective, Single-Arm, Phase II Study
Brief Title: Evaluating Nimotuzumab in Combination With AG Regimen for Pancreatic Cancer With Liver Metastases : A Prospective, Single-Arm, Phase II Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AG plus Nimotuzumab
Record Dates: First submitted 2024-05-05; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — nimotuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AG+nimotuzumab (Experimental): Pts with potentially resectable, treatment-naïve PCLM received nimotuzumab (400 mg, iv, d1, qw) and AG chemotherapy (gemcitabine 1000mg/m², Nab-paclitaxel 125mg/m², d1, d8, 21d cycle).
  Interventions: Drug: nimotuzumab; Drug: AG chemotherapy

INTERVENTIONS:
Drug: nimotuzumab — nimotuzumab (400 mg, iv, d1, qw)
Drug: AG chemotherapy — (gemcitabine 1000mg/m², Nab-paclitaxel 125mg/m², d1, d8, 21d cycle)

SUMMARY:
Patients with PCLM account for the majority of our department's pancreatic cancer cases and often have limited surgical options due to the aggressive nature of their tumors. For those with good performance status (ECOG PS 0-1), NCCN recommends gemcitabine + nab-paclitaxel (AG). Though nimotuzumab combined with gemcitabine improves survival, there remains scarce clinical data regarding its efficacy in conjunction with AG for treating PCLM. This study aims to evaluate the safety and efficacy of incorporating nimotuzumab with AG for PCLM.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age: 18-75 years old; 2) Physical strength KPS ≥ 60 points; 3) Pancreatic ductal epithelial adenocarcinoma with liver metastasis that has been diagnosed by pathological histology or cytology and is not suitable for radical radiotherapy or surgical treatment (should be at least 6 months away from the last adjuvant chemotherapy); 4) According to the RECIST 1.1 evaluation criteria, there should be at least one measurable and evaluable objective lesion (the longest diameter of the target lesion on spiral CT examination should be ≥ 10mm; if there is only lymph node metastasis, the shortest diameter should be ≥ 15mm); 5) Expected survival time ≥ 3 months; 6) Serum AST/ALT ≤ 5 times ULN; Total bilirubin ≤ 3 times ULN; Absolute count of granulocytes ≥ 1.5 × 109/L; Platelets ≥ 100 × 109/L; Hemoglobin ≥ 90 g/L; Creatinine clearance rate ≥ 60ml/min; 7) Voluntarily participate in this study, sign an informed consent form, and have good compliance; 8) Patients of childbearing age and their spouses are willing to take contraceptive measures.

Exclusion Criteria:

* 1) Prior to this study, the following treatments were received:

  1. Antitumor chemotherapy and molecular targeted therapy as a palliative measure
  2. The target lesion has undergone radiotherapy without any progression
  3. Within 4 weeks or currently participating in other therapeutic/intervention clinical trials 2) Received major surgery within 4 weeks; 3) Existing brain metastasis or leptomeningeal metastasis; 4) Have a history of other malignancies other than pancreatic cancer (except for cured cervical carcinoma in situ or skin basal cell carcinoma and other malignancies that have been cured for 5 years); 5) Merge symptomatic abdominal fluid that requires clinical treatment; 6) Accompanied by other serious illnesses, including but not limited to:

  <!-- -->

  1. Uncontrollable congestive heart failure (NYHA grade III or IV, see Appendix III), unstable angina, poorly controlled arrhythmias, uncontrolled moderate to high blood pressure (SBP>160mmHg or DBP>100mmHg)
  2. Active infection
  3. Difficult to control diabetes
  4. Mental illnesses that affect informed consent and/or adherence to protocols
  5. HIV infection
  6. There are serious illnesses that other researchers believe are not suitable for participating in this study 7) Known to be allergic to anti EGFR antibody preparations. 1.3 Exclusion criteria
* Failure to conduct effectiveness and/or safety evaluations; Serious violation of the protocol: While participating in this study, other chemotherapy drugs and/or modern Chinese medicine preparations with anti-cancer indications were used for treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
AEs | 3month
  Primary endpoints were adverse events (AEs),

SECONDARY OUTCOMES:
surgical conversion rates | 3month
  surgical conversion rates
R0 resection rates | 3month
  R0 resection rates
pathological complete response (pCR) rate | 3month
  pathological complete response (pCR) rate

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No